CLINICAL TRIAL: NCT01498107
Title: A Pilot Study Evaluating Engagement With a Platform Supporting Online Interventions for Common Mental Health Problems
Brief Title: Technology-enhanced Therapy: the SilverCloud Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridgeshire and Peterborough NHS Foundation Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Cecily Morrison, Research Associate, University of Cambridge
Allocation: Not Applicable | Model: Single Group | Purpose: Health Services Research
Other Study IDs: 609/M/C/791
Record Dates: First submitted 2011-12-14; First posted 2011-12-23 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Depression
Keywords: online intervention; computerized CBT; e-health
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: SilverCloud Platform — The SilverCloud online intervention will be provided as an alternative choice to paper manuals to support guided self-help for depression in a primary care mental health service. Participants will receive up to eight progress reviews on a weekly or fortnightly basis as agreed with their therapist with the intervention running not more than three months.

SUMMARY:
This pilot study investigates a new platform for supporting online interventions for common mental health problems called SilverCloud. It was developed from insights into interactive system design to address the problem of high attrition rates and poor engagement with online interventions. Through a range of methods, the study considers the role of four design strategies in engaging users in cognitive behavioural therapy. A service-based study, it concentrates on a clinical population with mild or moderate depression. Clinical outcome measures will be taken pre and post intervention use; demographic data of who did and did not choose the intervention collected, patterns of usage will be extracted from the log data and analysed; and qualitative interviews will be done to understand the relationship between patterns of usage and levels of engagement. The findings will be used to inform further developments of this and other online interventions and contribute to the development of methods for assessing online interventions.

The objectives of the pilot study are:

* To evaluate engagement with the online intervention in a realistic primary mental health care setting
* Assess engagement from multiple perspectives, including clinical efficacy and interaction design
* Contribute to further development of the online intervention
* Support preparation for a full-scale clinical trial

Research questions include:

* Does the online intervention decrease symptoms of depression?
* Who chooses to use the online intervention?
* What are the patterns of use of the online intervention?
* How successful are the four design principles, personal, interactive, supportive and social, in supporting engagement?

DETAILED DESCRIPTION:
INTERVENTION DESCRIPTION

SilverCloud platform SilverCloud is a platform on which to quickly build online interventions for common mental health problems. It utilises four design strategies that have been drawn from research in human-computer interaction: personal, interactive, supportive and social. SilverCloud is unusual among online interventions for its utilisation of current interactive design approaches.

* Personal: Users are encouraged to draw together all strands of the programme and build their own plan or "toolbox" for staying well and managing current and future mood difficulties.
* Interactive: Users can engage with the range of media, such as interactive quizzes, video presentation, online exercises and activities, homework, and mobile diary-keeping. These are meant to encourage reflection and personalization of the information.
* Supportive: Though mainly self-directed, each user in the programme will be assigned a therapist who will support them and provide feedback at specified intervals throughout the intervention on the activities that the user has chosen to share.
* Social: Users can gain a sense of other people using the system be seeing how many people liked an activity, or by sharing answers to an activity that are visible to all after moderation.

Mindbalance programme Mind Balance is a six-module programme built on the SilverCloud platform, incorporating psycho-educational and therapeutic elements of managing difficulties with low mood and depression. The programme draws primarily on the principles of cognitive behavioural therapy (CBT) and incorporates elements of mindfulness.

Service-based use The SilverCloud online intervention will be used as part of IAPT: Improving Access to Psychological Therapies. IAPT is a recent, centrally-developed, nationally- implemented, service model to implement National Institute for Clinical Excellent (NICE) guidelines for common mental health problems in primary care in the UK. It provides high throughput talking therapies at two levels of intensity to the adult population. The higher level provides therapy with a clinical psychologist and the lower level, guided self-help with a trained IAPT worker. The SilverCloud online intervention will be provided at the lower level of intensity as an alternative to manual-based guided self-help. Participants will receive up to eight reviews on a weekly or fortnightly basis as agreed with their IAPT worker with the intervention running not more than three months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depression with no co-morbidity of anxiety
* Appropriate for guided self-help in a primary care setting as determined by current IAPT procedures
* Owns a computer and has access to broadband internet
* Chooses to participate
* Gives consent to take part in the research

Exclusion Criteria:

* Are not comfortable reading in English
* Do not have adequate reading ability to use a guided self-help intervention
* Have had a CBT intervention within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Decrease in the Beck Depression Inventory Score | Change from baseline after 8 reviews have been completed in the online intervention

SECONDARY OUTCOMES:
Decrease in the Patient Health Questionnaire Score | Change from baseline after 8 reviews have been completed in the online intervention
Decrease in the Work and Social Adjustment Scale Score | Change from baseline after 8 reviews have been completed in the online intervention

CONTACTS AND LOCATIONS:
Overall Officials: Cecily Morrison, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Cambridgeshire Peterborough Foundation Trust: Improving Access to Psychological Therapies (IAPT), Cambridgeshire, Peterborough and Mid-Essex, United Kingdom